CLINICAL TRIAL: NCT03213990
Title: A Phase III Randomised Controlled Trial of Continuous Beta-lactam Infusion Compared With Intermittent Beta-lactam Dosing in Critically Ill Patients
Brief Title: Beta-Lactam InfusioN Group Study
Acronym: BLING III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGI-CCT254643
Record Dates: First submitted 2017-06-05; First posted 2017-07-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Sepsis
Keywords: Sepsis; Beta-lactam antibiotics
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Infusion (Other): The prescribed Beta-lactam is administered by a continuous infusion.
  Interventions: Other: Continuous infusion
- Intermittent infusion (Other): the prescribed Beta-lactam is administered by intermittent infusion over 30 minutes
  Interventions: Other: Intermittent infusion

INTERVENTIONS:
Other: Continuous infusion — Clinician prescribed beta-lactam antibiotic will be administered via continuous infusion for as long as prescribed whilst in the ICU
  Arms: Continuous Infusion
Other: Intermittent infusion — Clinician prescribed beta-lactam antibiotic will be administered via intermittent infusion for as long as prescribed whilst in the ICU
  Arms: Intermittent infusion

SUMMARY:
The purpose of this study is to find out whether continuous infusion of beta-lactam antibiotics or intermittent infusion or beta-lactam antibiotics, offers more health advantages to patients or if there is no difference.

The investigators will be looking to see whether patients receiving beta-lactams via one administration method or the other have a better chance of recovering from their illness. They will also be looking at long term outcomes such as quality-of-life and healthcare resource use.

Sepsis is caused by toxic substances (toxins) from bacteria and other organism entering the bloodstream from a site of infection. In some people, the infection can progress to sepsis and septic shock where the functions of organs in the body are affected. Patients suffering from sepsis and septic shock are commonly managed in the intensive care unit (ICU) where they are prescribed antibiotics as standard therapy, as well as other therapies to support the functions of the body.

Beta-lactam antibiotics are a group of antibiotics commonly used to treat infection in patients with sepsis and septic shock.

Currently, beta-lactam antibiotics are most commonly given to patients be intermittent infusions, that is, given at regular intervals throughout 24 hours. New research suggests that giving beta-lactam antibiotics as a continuous infusion may mean that antibiotic concentrations in the blood remain more consistent and may be more effective at killing bacteria.

However, the benefit to the patient by giving beta-lactams via continuous infusion has not been tested in a high-quality, large clinical trial.

DETAILED DESCRIPTION:
Aim To conduct a multicentre randomised, controlled trial (RCT) to determine whether continuous infusion of a beta-lactam antibiotic (piperacillin-tazobactam or meropenem) results in decreased all cause Day 90 mortality compared with intermittent beta-lactam antibiotic infusion in critically ill patients with sepsis.

Hypothesis The BLING III Study will test the hypothesis that patients managed in the ICU with sepsis, the administration of beta-lactam antibiotics via continuous infusion decreases Day 90 mortality compared with intermittent infusion Design This BLING III study is a prospective, multicentre, open, phase III, RCT. Participants commenced on one of two beta-lactam antibiotics (piperacillin-tazobactam or meropenem) will be randomised to receive the beta-lactam antibiotic via either continuous infusion or intermittent infusion over 30 minutes for the treatment course while in the ICU for up to 90 days after randomisation. For participants where the beta-lactam antibiotic is subsequently changed from piperacillin-tazobactam to meropenem or vice versa for ongoing treatment of the infectious episode, the new prescription will continue to be administered in the allocated method (continuous infusion or intermittent infusion over 30 minutes).

Permuted block randomisation with variable block sizes and stratified by site will be conducted via a password-protected, secure web-based interface.

The primary endpoint for this trial will be death from all causes at 90 days.

7,000 patients will be enrolled into this study from approximately 70 ICUs worldwide, with approximately 35 ICUs in Australian and New Zealand hospitals.

For eligible patients, the administration method of beta-lactam antibiotic, either piperacillin-tazobactam or meropenem, will be randomised to either continuous infusion or intermittent infusion over 30 minutes. The choice of beta-lactam antibiotic and the dose and dosing interval (i.e. the dose the patient will receive in 24 hours) will be determined by the treating physician prior to randomisation.

For all patients, data will be collected at baseline and daily whilst in the ICU. Patients will be followed up to day 14, regardless of location in the hospital, to determine test of cure and to identify new acquisition, colonisation or infection with an multi-resistant organism. Additional follow up will occur at 90 days post randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Documented site of infection or strong suspicion of infection
2. At the time of the assessment of suitability for the study, the treating physician expects the patient will require treatment in the ICU that extends beyond the next calendar day
3. The treating physician has chosen piperacillin-tazobactam or meropenem to treat the episode of infection
4. The treating physician is uncertain if administration of the chosen antibiotic by intermittent or continuous infusion is superior
5. One or more organ dysfunction entry criteria in the previous 24 hours

   * i. Mean arterial pressure < 60 mmHg for at least 1 hour
   * ii. Vasopressors required for > 4 hours
   * iii. Respiratory support using supplemental high flow nasal prongs, continuous positive airway pressure, bilevel positive airway pressure or invasive mechanical ventilation for at least 1 hour
   * iv. Serum creatinine concentration > 220 µmol/L

Exclusion Criteria:

1. Age less than 18 years
2. Receipt of piperacillin-tazobactam or meropenem for more than 24 hours during current infectious episode
3. Patients who are known or suspected to be pregnant
4. Patient has a known allergy to piperacillin-tazobactam or meropenem or penicillin
5. Receiving renal replacement therapy at the time of assessment for eligibility
6. The treating physician is not committed to provision of advanced life-support, including mechanical ventilation, dialysis and vasopressor administration, for at least the next 48 hours
7. Death is deemed imminent and inevitable
8. The patient has previously been enrolled in BLING III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7203 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 90 Days after randomisation
  Patient mortality status assessed at 90 days after randomisation

SECONDARY OUTCOMES:
Clinical Cure | Day 14 post randomisation
  Clinical cure will be defined as the completion of the beta-lactam antibiotic treatment course (on or prior to Day 14) without recommencement of antibiotic therapy within 48 hours of cessation.
  Participants discharged from hospital within 14 days following randomisation will be considered to meet the definition of clinical cure. Participants who decease while receiving the antibiotic treatment course or where antibiotic therapy is ceased in the setting of death being deemed imminent and inevitable, will be assessed as not meeting the criteria for clinical cure.
New acquisition, colonisation or infection | up to 14 days post randomisation or hospital discharge, whichever is sooner
  New acquisition, colonisation or infection with an Multi-resistant organism (MRO) or Clostridium difficile diarrhoea
All cause ICU mortality | up to 90 days
  Patient mortality status assessed at ICU discharge
All cause hospital mortality | up to 90 days
  Patient mortality status assessed at hospital discharge

OTHER OUTCOMES:
ICU length of stay | up to 90 days
  Patient assessment of time spent in the ICU
Hospital length of stay | up to 90 days
  Patient assessment of time spent in hospital.
Quality of life | 90 days after randomisation
  Quality of life measured with the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L)
Health services use | up to 90 days after randomisation
  Additional follow up at Day 90 for the purpose of economic evaluation will be conducted for Australian, New Zealand and sites from participating regions only. Follow up at Day 90 will include recording readmission to hospital and ICU within 90 days and will assess quality of life and functional capacity using the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) questionnaire (if not deceased).38 The consent document used at participating sites will detail the inclusion of a quality of life questionnaire at Day 90.
Cost effectiveness analysis | up to 90 days
  A cost-effectiveness analysis at 90 days following randomisation will be conducted as a nested cohort in Australian, New Zealand and other potential regional sites. Cost data will be derived from health care utilisation to Day 90, estimated through standard per diem ICU and hospital costs. The analysis will be conducted from a health care payer perspective, comparing health care utilisation costs and quality-adjusted life years gained (measured by the EQ-5D-5L) between treatment arms. Where feasible, the cost-effectiveness analysis will be conducted in other country-specific regions. Depending on the outcome from the primary trial, several further analyses are planned including a longer-term cohort study and a modelled economic evaluation. The BLING III cost-effectiveness analysis will be informed by a separate Statistical Analysis Plan.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lipman, Study Chair — The George Institute
Locations (103):
- Australia (25):
  - Bankstown Hospital, Bankstown, New South Wales
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincents Hosptial, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Darwin Hospital, Casuarina, Northern Territory
  - The Wesley Hospital, Auchenflower, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Caboolture Hospital, Caboolture, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Hospital, Bendigo, Victoria
  - Box Hill Hospital - Eastern Health, Box Hill, Victoria
  - Geelong University Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Belgium (8):
  - Hôpital Erasme, Brussels, Anderlecht
  - ZNA Stuivenberg, Antwerp
  - Universitair ziekenhuis Antwerpen, Antwerp
  - Universitair ziekenhuis Brussel, Brussels
  - Civil Hospital Marie Curie, Charleroi
  - Maria Middelares, Ghent
  - Universitair ziekenhuis Gent, Ghent
  - Clinique Saint Pierre, Ottignies
- France (5):
  - Ch Salon de Provence, Salon-de-Provence, Bouche Du Rhone
  - Nimes University Hospital, Nîmes, Nimes
  - Centre Hospitalier Henri Duffaut, Avignon, Vaucluse
  - Brabois, Nancy
  - Poitiers University Hospital, Poitiers
- Malaysia (2):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Selangor
- New Zealand (6):
  - Auckland City Hospital - CVICU, Auckland
  - Auckland City Hospital - DCCM, Auckland
  - Middlmore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- Sweden (3):
  - Helsingborg Hospital, Helsingborg
  - Skane Lund University Hospital, Lund
  - Skane University Malmo Hospital, Malmo
- United Kingdom (54):
  - Royal Berkshire Hospital, Reading, Berkshire
  - Kings College Hospital, London, Brixton
  - Princess Royal University Hospital, Orpington, Bromley
  - Stoke Mandeville Hospital, Aylesbury, Buckinghamshire
  - Milton Keynes University Hospital, Milton Keynes, Buckinghamshire
  - Countess of Chester Hospital, Chester, Cheshire
  - Dorset County Hospital, Dorchester, Dorset
  - Poole Hospital, Poole, Dorset
  - University Hospital of North Tees, Stockton-on-Tees, Durham
  - Ipswich Hospital, Ipswich, East Suffolk
  - Darent Valley Hospital, Dartford, England
  - Maidstone Hospital, Maidstone, England
  - Derriford Hospital, Plymouth, England
  - Broomfield Hospital, Chelmsford, Essex
  - Golden Jubilee National Hospital, Clydebank, Glasgow
  - Royal Bolton Hospital, Bolton, Greater Manchester
  - Charing Cross Hospital, London, Hammersmith
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Southampton General Hospital, Southampton, Hampshire
  - Royal Hampshire County Hospital, Winchester, Hampshire
  - Hereford County Hospital, Hereford, Herefordshire
  - Watford General Hospital, Watford, Hertfordshire
  - Medway Maritime Hospital, Gillingham, Kent
  - Kingston Hospital, Kingston upon Thames, Kent
  - Tunbridge Wells Hospital, Royal Tunbridge Wells, Kent
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - The Royal Marsden, Chelsea, London
  - Guy's & St Thomas' Hospital London, Lambeth, London
  - St Georges Hospital, Tooting, London
  - The Royal London Hospital, Whitechapel, London
  - Royal Victoria Infirmary, Newcastle, Northhumberland
  - Newcastle Freeman Hospital, Newcastle, Northumberland
  - The Queens Medical Centre, Nottingham, Nottinghamshire
  - Kingsmill Hospital, Sutton in Ashfield, Nottinghamshire
  - St Marys Hospital, London, Paddington
  - Whiston Hospital, Rainhill, Prescot
  - Hammersmith Hospital, London, Shepherds Bush
  - James Cook University Hospital South Tees, Middlesbrough, South Tees
  - Frimley Park Hospital, Frimley, Surrey
  - Royal Surrey County Hospital, Guildford, Surrey
  - Sunderland Royal Hospital, Sunderland, Tyne and Wear
  - University Hospital of Wales, Cardiff, Wales
  - University Hospital Coventry & Warwickshire, Coventry, Warwickshire
  - Queen Elizabeth Medical Centre, Birmingham, West Midlands
  - Pinderfields General Hospital, Wakefield, West Yorkshire
  - Bristol Royal Infirmary, Bristol
  - Northumbria Specialist Emergency Hospital, Cramlington
  - Ninewells Hospital, Dundee
  - Glasgow Royal Infirmary, Glasgow
  - Hull Royal Infirmary, Hull
  - Whittington Health, London
  - Queen's Hospital, Romford
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Undecided
Yet to be decided

REFERENCES:
- [Derived] Dulhunty JM, Brett SJ, De Waele JJ, Rajbhandari D, Billot L, Cotta MO, Davis JS, Finfer S, Hammond NE, Knowles S, Liu X, McGuinness S, Mysore J, Paterson DL, Peake S, Rhodes A, Roberts JA, Roger C, Shirwadkar C, Starr T, Taylor C, Myburgh JA, Lipman J; BLING III Study Investigators. Continuous vs Intermittent beta-Lactam Antibiotic Infusions in Critically Ill Patients With Sepsis: The BLING III Randomized Clinical Trial. JAMA. 2024 Aug 27;332(8):629-637. doi: 10.1001/jama.2024.9779. PMID 38864155
- [Derived] Lipman J, Brett SJ, De Waele JJ, Cotta MO, Davis JS, Finfer S, Glass P, Knowles S, McGuinness S, Myburgh J, Paterson DL, Peake S, Rajbhandari D, Rhodes A, Roberts JA, Shirwadkar C, Starr T, Taylor C, Billot L, Dulhunty JM. A protocol for a phase 3 multicentre randomised controlled trial of continuous versus intermittent beta-lactam antibiotic infusion in critically ill patients with sepsis: BLING III. Crit Care Resusc. 2019 Mar;21(1):63-68. PMID 30857514

DOCUMENTS (3):
  • Study Protocol: PKPD Substudy (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03213990/Prot_000.pdf
  • Study Protocol: BLING III PKPD substudy protocol (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03213990/Prot_002.pdf
  • Statistical Analysis Plan (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03213990/SAP_001.pdf